CLINICAL TRIAL: NCT04516577
Title: Severity of Patients With Pulmonary Alveolar Proteinosis (PAP) Through Disease Severity Score (DSS), Severity and Prognosis Score of PAP (SPSP) and SPSPII
Brief Title: Updated Severity and Prognosis Score of Pulmonary Alveolar Proteinosis
Status: Completed | Type: Observational
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Jin-Fu Xu, Chief of Respiratory and Critical Care Medicine, Shanghai Pulmonary Hospital, Shanghai, China
Other Study IDs: 2020073195
Record Dates: First submitted 2020-08-11; First posted 2020-08-18 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: Pulmonary Alveolar Proteinosis
MeSH Terms: conditions — Pulmonary Alveolar Proteinosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Shanghai Pulmonary Hospital: Shanghai Pulmonary Hospital is a hospital specializing in the treatment of lung diseases. Many patients with pulmonary alveolar proteinosis receive treatment in this hospital.
  Interventions: Other: Assesssing the severity of pulmonary alveolar proteinosis
- Peking Union Medical College Hospital: Peking Union Medical College Hospital is a famous hospital in China. Many patients with rare pulmonary disease receive treatment in this hospital.
  Interventions: Other: Assesssing the severity of pulmonary alveolar proteinosis
- Nanjing Drum Tower Hospital: The Department of Respiratory and Critical Care Medicine of Nanjing Drum Tower Hospital has been focusing on the research of rare pulmonary diseases for many years.

INTERVENTIONS:
Other: Assesssing the severity of pulmonary alveolar proteinosis — Three severity scores will be used to assess the severity of patients with pulmonary alveolar proteinosis.
  Groups: Peking Union Medical College Hospital; Shanghai Pulmonary Hospital

SUMMARY:
By updating the chest HRCT scoring criteria of patients with pulmonary alveolar proteinosis, a new and more perfect system for evaluating the severity of alveolar proteinosis will be established.

DETAILED DESCRIPTION:
In past, investigators summarized a method that was the severity and prognosis of pulmonary alveolar proteinosis (SPSP) to assess the severity and prognosis of patients with autoimmune pulmonary alveolar proteinosis (auto PAP). The SPSP included five aspects: smoking, symptom, PaO2, chest CT score at specific levels (aortic arch, carina, pulmonary vein confluence, and superior septal level) and DLCO %predicted. But the chest CT score only focused on range of lesions, and inaccurate. So, investigators plan to adopt new score which involves the assessing to range and density.

In the new Chest HRCT score, we added the density score. The average density of the lesions at a particular level of the patient's chest HRCT was measured by computer and classified into three degrees: mild (less than -400), moderate (greater than -400 and less than -100) and severe (greater than 100), denoted as 1 ', 2 'and3', respectively.

The range score of lung opacity was estimated using a five-point scale: no opacity = 0; opacity involving < 25% of a region of hemithorax = 1; 25-50% = 2; 50-75% = 3; and ≥ 75% = 4.

The lesion score for each layer is equal to the density score multiplied by the range score. The chest HRCT score was calculated by summing the lung opacity scores of the four representative regions of each hemithorax, and divided into several level: no opacity = 0; ≤10 = 1; 11 - 20 = 2; 21 - 30 = 3; 31 -40 = 4; > 40 = 5.

According to the new chest HRCT score, the SPSP will be updated to SPSP II. In this study, patients with auto PAP from three centers (Shanghai Lung Hospital, Peking Union Medical College Hospital and Nanjing Drum Tower Hospital) were enrolled to evaluate the severity of disease severity score (DSS), SPSP and SPSP II, respectively, to evaluate the pros and cons of different scores and their impact on prognosis.

About 30 newly diagnosed auto PAP patients were recruited, and were assess disease severity on the basis on SPSP II scores. According to SPSP II scores, appropriate treatment was used for the patients, who were followed up for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* The patients had be diagnosed with autoimmune pulmonary alveolar proteinosis through pathology or bronchial alveolar lavage fluid (BALF).
* The patients are old than 18 year.
* .Every patient had a complete medical history, chest HRCT, pulmonary function and arterial blood gas analysis.
* The patients have high level antibody of GM-CSF in serum or BALF.

Exclusion Criteria:

* The patients had a congenital or secondary pulmonary alveolar proteinosis.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The patients had be diagnosed with autoimmune pulmonary alveolar proteinosis. Every patient had a complete medical history, chest HRCT, pulmonary function and arterial blood gas analysis.
Sampling Method: Probability Sample
Enrollment: 231 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
The severity and prognosis of pulmonary alveolar proteinosis | From July 2020 to December 2021
  The second severity and prognosis score of PAP (SPSP II) involves the range and density of lesion in chest CT of patients

CONTACTS AND LOCATIONS:
Overall Officials: Xinlun Tian, Dr, Principal Investigator — Peking Union Medical College Hospital; Yonglong Xiao, Dr, Principal Investigator — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Locations (1):
- Shanghai pulmonary hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bai JW, Huang JN, Shi SY, Ge A, Lu HW, Sun XL, Gu SY, Liang S, Cheng KB, Tian XL, Xiao YL, Xu KF, Xu JF. Updated severity and prognosis score of pulmonary alveolar proteinosis: A multi-center cohort study in China. Front Med (Lausanne). 2023 Feb 7;10:1058001. doi: 10.3389/fmed.2023.1058001. eCollection 2023. PMID 36824611